CLINICAL TRIAL: NCT02080195
Title: A Phase I/II Study of Nonmyeloablative Conditioning and Transplantation of Human Leukocyte Antigen (HLA)-Matched, Partially HLA-mismatched, HLA-haploidentical or Matched Unrelated Bone Marrow for Patients With Refractory SLE
Brief Title: Nonmyeloablative Conditioning and Transplantation for Patients With Refractory Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was unable to accrue subjects
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Stem Cell Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J13134; NA_00082453 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Lupus Erythematosus; Graft-versus-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Tacrolimus; Mycophenolic Acid; thymoglobulin; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nonmyeloablative Conditioning and BMT (Experimental): Nonmyeloablative conditioning with rabbit antithymocyte globulin, cyclophosphamide, fludarabine, and total body irradiation. Allogeneic bone marrow transplant on Day 0. Graft versus host disease (GVHD) prophylaxis with cyclophosphamide, mycophenolate mofetil, and tacrolimus.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Rabbit antithymocyte globulin; Radiation: Total body irradiation; Biological: Allogeneic bone marrow transplant

INTERVENTIONS:
Drug: Cyclophosphamide — 14.5 mg/kg/day on Days -6 and -5. 50 mg/kg/day on Days 3 and 4.
  Other Names: Cytoxan; Cy
Drug: Fludarabine — 30 mg/m^2/day on Days -6 through -2.
  Other Names: Fludara
Drug: Tacrolimus — Starting on Day 5. Dose will be adjusted according to blood levels.
  Other Names: FK-506; Prograf
Drug: Mycophenolate Mofetil — 15 mg/kg three times per day from Day 5 to Day 35.
  Other Names: Cellcept; MMF
Drug: Rabbit antithymocyte globulin — 0.5 mg/kg on Day -9. 2 mg/kg/day on Days -8 and -7.
  Other Names: Thymoglobulin
Radiation: Total body irradiation — 200 centigray on Day -1.
Biological: Allogeneic bone marrow transplant — Infusion on Day 0.
  Other Names: BMT

SUMMARY:
The main goal of the study is to determine if bone marrow transplant (BMT) from a less specific pool of donors in combination with high dose cyclophosphamide can induce remission of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a devastating systemic autoimmune disease that predominantly affects young women, is more common in African-Americans than in whites, and results in poor quality of life. Lupus has no cure, and up to 90% of patients require corticosteroids for disease control. More than half of patients with lupus have permanent organ damage, much of which is either directly due to or increased by corticosteroids. To satisfactorily manage moderate-to-severe SLE, the investigators need effective treatments that will allow corticosteroid-sparing.

High-dose chemotherapy followed by autologous BMT or peripheral blood progenitor transplantation (PBSCT) has been proposed as a novel approach to treat severe autoimmune diseases. Allogeneic BMT is not currently utilized for the routine treatment of SLE because of the significant morbidity (GVHD) and mortality associated with the procedure.

The investigators have recently developed an approach to BMT using post-transplant cyclophosphamide that allows us to safely perform allogeneic BMT from matched, mismatched, unrelated or haploidentical donors. Transplant-related mortality, graft-failure and risk of GVHD have been very low with this approach. Furthermore, this approach allows us to greatly expand the donor pool since any patient shares exactly one HLA haplotype with each biological parent or child and half of siblings, an eligible haploidentical donor can be identified rapidly in nearly all cases.

This trial will employ a fludarabine + cyclophosphamide conditioning along with posttransplantation cyclophosphamide on for patients with refractory SLE. The purpose of this trial is to improve the salvage rate for patients with refractory SLE through a reformatting of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Four or more American College of Rheumatology (ACR) criteria for the classification of SLE or 4 or more of the SLICE criteria
* Involvement of one or more of the following organ systems: renal, neurologic, hematologic, cardiac, pulmonary, gastrointestinal
* A lack of response to corticosteroids in moderate-to-high doses, and to either an equivalent degree of immunosuppression with azathioprine, methotrexate, cyclosporin, tacrolimus, belimumab, rituximab, mycophenolate mofetil, and/or appropriate other treatment
* Patients should be eligible for transplantation according to the BMT Policy Manual

Exclusion Criteria:

* Age less than 18 years and over 75 years
* Any risk of pregnancy
* Patients who are preterminal or moribund

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bolaños-Meade, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonmyeloablative Conditioning and BMT: Nonmyeloablative Conditioning and Bone Marrow Transplant in Systemic Lupus Erythematosus patients
  Cyclophosphamide: Cyclophosphamide (alkylating agent) conditioning regimen and post transplantation cyclophosphamide with matched, partially matched, haplo-identical or unrelated donors
  Sodium-2-mercapto ethane sulphonate: Antineoplastic detoxifying agent
  Fludarabine monophosphate: Purine antimetabolite
  Tacrolimus: Calcineurin inhibitor
  Mofetil: Immunosuppressant
  Rabbit antithymocyte globulin: Selective immunosuppressant
Period: Overall Study
Arm/Group | Nonmyeloablative Conditioning and BMT
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of the Conditioning Regimen and Post Transplantation Cyclophosphamide in Refractory SLE Patients With Donors Having Various Degrees of Matching
Description: Number of participants who were alive at 1 year after transplant and who had not suffered graft rejection, acute or chronic GVHD, or Grade 3 or higher (CTCAE V4.0) adverse events.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: RIFLE Score
Description: Change in Responder Index for Systemic Lupus Erythematosis (RIFLE) assessment. This is a qualitative assessment of organ function. The 12 month response will be assessed as:
  complete= complete or partial resolution in more than one organ, partial= complete or partial resolution in at least one organ, the same= no change or no worsening in any organ, worse= worsening in any organ
Time Frame: 1 year
Population: The only enrolled participant on this study was never assessed for a follow-up RIFLE scale, so no data was collected for this outcome measure.
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival
Description: Number of patients alive and alive without relapse, respectively.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Participants
  Overall Survival | 1
  Event Free Survival | 1

4. Secondary Outcome: Graft Failure
Description: Number of participants with primary and/or secondary graft failure.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Participants
  Primary graft failure | 0
  Secondary graft failure | 0

5. Secondary Outcome: Acute Graft Versus Host Disease (GVHD)
Description: Percentage of participants who developed grades II-IV and grades III-IV acute GVHD. Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Participants
  Grades II-IV acute GVHD | 0
  Grades III-IV acute GVHD | 0

6. Secondary Outcome: Chronic Graft Versus Host Disease (GVHD)
Description: Percentage of participants who developed chronic GVHD as defined by the NIH consensus criteria. This system gives scores from 0 to 3 for Karnofsky performance score, skin, mouth, eyes, gastrointestinal, liver, lungs, joints, and genitals, as well as an overall severity (mild, moderate, or severe).
  Mild chronic GVHD involves only 1 or 2 organs or sites (except the lung), with no clinically significant functional impairment (maximum of score 1 in all affected organs or sites).
  Moderate chronic GVHD involves 1) at least 1 organ or site with clinically significant but no major disability (maximum score of 2 in any affected organ or site) OR 2) 3 or more organs or sites with no clinically significant functional impairment (maximum score of 1 in all affected organs or sites).
  Severe chronic GVHD indicates major disability caused by chronic GVHD (score of 3 in any organ or site).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nonmyeloablative Conditioning and BMT
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed weekly through at least Day 60.
Description: Reportable serious adverse events per protocol include: any mortality within the first 100 days after bone marrow transplant (BMT), any graft failures (defined as <5% donor chimerism) associated with failure of neutrophil recovery to >500/mm³ by day ~60 after transplantation, and all unexpected events as deemed significant by the PIs. Other events were neither tracked nor reported for this study.
Arm/Group | Nonmyeloablative Conditioning and BMT
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT02080195/Prot_SAP_000.pdf